CLINICAL TRIAL: NCT06307002
Title: Evaluating the Impact of a Contraception Education Game: What's My Method? on Contraceptive Self-efficacy and Clinical Outcomes in Barbados
Brief Title: Evaluating What's My Method? in Barbados
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Quinnipiac University (Other)
Collaborators: Barbados Family Planning Association (Unknown)
Responsible Party: Principal Investigator, Elena Bertozzi, Professor, Director of Game Design & Development, Quinnipiac University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CAS_EB_2024
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Contraception Behavior
Keywords: Contraceptive Self-efficacy; Reproductive Empowerment; Videogame
MeSH Terms: conditions — Contraception Behavior

STUDY DESIGN:
Intervention Model Description: This is a 2 arm randomized controlled trial comparing standard of care (SOC) counseling alone to What's My Method? (WMM) gameplay in addition to SOC.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (No Intervention): The control group will receive SOC counseling, defined as the current practice at our partner institutions. Patients presenting for contraceptive counseling are given informational pamphlets and have the option to review additional materials posted on the clinic walls and on a rotating slide deck on a digital screen. During their counseling session with a provider, they review eligible methods and can make a decision about whether or not to adopt a method, and to select and initiate the contraception of their choice.
- WMM Arm (Experimental): The intervention group will be provided with a tablet loaded with the WMM game which will be played in the waiting room prior to their visit. They will then receive SOC counseling, defined as the current practice at our partner institutions. Patients presenting for contraceptive counseling are given informational pamphlets and have the option to review additional materials posted on the clinic walls and on a rotating slide deck on a digital screen. During their counseling session with a provider, they review eligible methods and can make a decision about whether or not to adopt a method, and to select and initiate the contraception of their choice.
  Interventions: Other: Playing a contraception education videogame

INTERVENTIONS:
Other: Playing a contraception education videogame — The WMM game is divided into three parts- a reproductive anatomy quiz ("Parts"), an interactive tool for education about each individual birth control method ("Methods"), and a section in which players help avatar couples choose the most effective method for them.
  Arms: WMM Arm

SUMMARY:
The purpose of this study is to measure the impact of the What's My Method game on participants' sense of agency, education, and empowerment around contraceptive decision-making. Patients receiving standard of care contraceptive counseling will be compared to those who play the game in addition to counseling.

DETAILED DESCRIPTION:
Contraceptive self-care has been identified by the WHO as critical to achieving milestones for female empowerment and well-being. This focus reflects a shift in global public health attitudes regarding contraceptive provision from a top-down approach, where childbearing persons receive directives from medical providers, towards an approach that encourages self-determination and individual agency. Implementing contraceptive counseling and education through the lens of reproductive empowerment requires that the focus of the intervention be on the childbearing persons and their needs. There is a clear need for improvement in contraceptive counseling in Barbados. As per the United Nations dashboard, the modern contraceptive prevalence rate is 49% and providers report that abortion is often used as birth control.

Digital health interventions have been validated as successful high-impact practices to support healthy reproductive behaviors. These interventions include SMS campaigns , artificial intelligence-based chatbots, and interactive websites which provide information and offer tools to help choose appropriate methods. These studies demonstrate that digital media are an effective way to reach the target audience and communicate information about reproductive health. Barbadian clinics have not yet integrated digital technology to support CC; they rely on pamphlets and posters for information dissemination.

This study seeks assess the impact of supplementing SOC counseling with a digital game that provides detailed information about family planning methods, their benefits and side effects. The information is communicated through using animations and images and reinforced through experimentation and context.

ELIGIBILITY:
Inclusion Criteria:

* - English-speaking
* Capable of using a tablet
* Childbearing individuals
* Individuals/Couples seeking family planning counseling (one response collected per couple)

Exclusion Criteria:

* Unable to provide informed consent due to intellectual or physical impairment - Under the age of 18 unless accompanied by a parent

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Persons who can become pregnant
Enrollment: 70 (Actual)
Dates: Start 2024-03-11 (Actual); Primary Completion 2024-11-13 (Actual); Study Completion 2024-11-13 (Actual)

PRIMARY OUTCOMES:
Contraceptive Self-Efficacy (CSE) score | 30-70 minutes
  Participants will complete a survey after their contraceptive counseling appointment

SECONDARY OUTCOMES:
Method Adoption | 30-70 minutes
  Participant will indicate if they desire a method and obtain or request an appointment to obtain said method
Qualitative feedback on game intervention | 50-90 minutes
  Group that played the game will complete 4 question assessment of experience

CONTACTS AND LOCATIONS:
Locations (1):
- Barbados Family Planning Association, Bridgetown, Saint Michaels, Barbados

IPD SHARING:
Plan to Share IPD: Yes
Participant identifying information will not be collected as part of the study. Study data (scores on surveys, rate of method adoption) will be posted on a publicly available shared repository for use by other researchers.
Supporting Information: CSR, Analytic Code
Time Frame: within 3 months of publication.
Access Criteria: Data already collected is available at the Center for Open Science
URL: https://osf.io/q2w6u/?view_only=9c0b192d05b34c73b7ccf34347f79947

REFERENCES:
- [Background] Bearak JM, Popinchalk A, Beavin C, Ganatra B, Moller AB, Tuncalp O, Alkema L. Country-specific estimates of unintended pregnancy and abortion incidence: a global comparative analysis of levels in 2015-2019. BMJ Glob Health. 2022 Mar;7(3):e007151. doi: 10.1136/bmjgh-2021-007151. PMID 35332057
- [Background] Bertozzi E, Bertozzi-Villa A, Kulkarni P, Sridhar A. Collecting family planning intentions and providing reproductive health information using a tablet-based video game in India. Gates Open Res. 2018 Sep 7;2:20. doi: 10.12688/gatesopenres.12818.2. eCollection 2018. PMID 29984358
- [Background] Chukwu E, Gilroy S, Addaquay K, Jones NN, Karimu VG, Garg L, Dickson KE. Formative Study of Mobile Phone Use for Family Planning Among Young People in Sierra Leone: Global Systematic Survey. JMIR Form Res. 2021 Nov 12;5(11):e23874. doi: 10.2196/23874. PMID 34766908
- [Background] Dehlendorf C, Fitzpatrick J, Fox E, Holt K, Vittinghoff E, Reed R, Campora MP, Sokoloff A, Kuppermann M. Cluster randomized trial of a patient-centered contraceptive decision support tool, My Birth Control. Am J Obstet Gynecol. 2019 Jun;220(6):565.e1-565.e12. doi: 10.1016/j.ajog.2019.02.015. Epub 2019 Feb 11. PMID 30763545
- [Background] Fiellin LE, Hieftje KD, Pendergrass TM, Kyriakides TC, Duncan LR, Dziura JD, Sawyer BG, Mayes L, Crusto CA, Forsyth BW, Fiellin DA. Video Game Intervention for Sexual Risk Reduction in Minority Adolescents: Randomized Controlled Trial. J Med Internet Res. 2017 Sep 18;19(9):e314. doi: 10.2196/jmir.8148. PMID 28923788
- [Background] Hamidi OP, Deimling T, Lehman E, Weisman C, Chuang C. High Self-Efficacy Is Associated with Prescription Contraceptive Use. Womens Health Issues. 2018 Nov-Dec;28(6):509-513. doi: 10.1016/j.whi.2018.04.006. Epub 2018 Aug 18. PMID 30131220
- [Background] Stephenson J, Bailey JV, Gubijev A, D'Souza P, Oliver S, Blandford A, Hunter R, Shawe J, Rait G, Brima N, Copas A. An interactive website for informed contraception choice: randomised evaluation of Contraception Choices. Digit Health. 2020 Jun 26;6:2055207620936435. doi: 10.1177/2055207620936435. eCollection 2020 Jan-Dec. PMID 32704380
- [Background] Laidlaw R, Dixon D, Morse T, Beattie TK, Kumwenda S, Mpemberera G. Using participatory methods to design an mHealth intervention for a low income country, a case study in Chikwawa, Malawi. BMC Med Inform Decis Mak. 2017 Jul 5;17(1):98. doi: 10.1186/s12911-017-0485-6. PMID 28679428
- [Background] Lepore C, McNamara M, Miclette K, Vash-Margita A. Assessment of a Novel Interactive Website to Inform Adolescent and Young Adult Decision-Making about Contraception. J Pediatr Adolesc Gynecol. 2024 Apr;37(2):149-155. doi: 10.1016/j.jpag.2023.10.006. Epub 2023 Nov 6. PMID 37935279
- [Background] Wang H, Gupta S, Singhal A, Muttreja P, Singh S, Sharma P, Piterova A. An Artificial Intelligence Chatbot for Young People's Sexual and Reproductive Health in India (SnehAI): Instrumental Case Study. J Med Internet Res. 2022 Jan 3;24(1):e29969. doi: 10.2196/29969. PMID 34982034
- [Background] Whiting-Collins L, Grenier L, Winch PJ, Tsui A, Donohue PK. Measuring contraceptive self-efficacy in sub-Saharan Africa: development and validation of the CSESSA scale in Kenya and Nigeria. Contracept X. 2020 Oct 9;2:100041. doi: 10.1016/j.conx.2020.100041. eCollection 2020. PMID 33145490